CLINICAL TRIAL: NCT05543772
Title: Evaluation of Blood Sampling From a Pre-existed Peripheral Intravenous Catheter Line (Indwelling Line): a Technique to Keep Optimal Specimen After Fluid Flush
Brief Title: Evaluation of Blood Sampling From a Pre-existed Peripheral Intravenous Catheter Line
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Dunya N Alfaraj, MD, Emergency Consultant, Imam Abdulrahman Bin Faisal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IABFUniversity
Record Dates: First submitted 2022-06-05; First posted 2022-09-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies | interventions — Saline Solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Normal saline (Experimental): Study will be held in King Fahad University Hospital during a year after obtaining the IRB approval. Selection of study participants will be depending on their health status and the investigators will exclude pediatric participants. Two blood samples will be collected from participants. First one is after the insertion of the intravenous peripheral line. The second is after fluid infusion through the same line. Samples will be sent to the laboratory then. Results will be collected and analyzed.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — participant will be given 500 ml normal saline through intravenous access. blood sample will be extracted before and after giving normal saline using same intravenous catheter

SUMMARY:
Background: Peripheral Intravenous catheter (PIVC) is a frequently used device for intravascular access. It is usually indicated to administer intravenous fluid and medications. However, the investigators could possibly utilize this line for blood sampling even after using it as a fluid port.

DETAILED DESCRIPTION:
Aims: To investigate the quality of previously flushed PIVC sample and the effectiveness of the withdrawal technique.

Methodology: Study will be held in King Fahad University Hospital during a year after obtaining the IRB approval. Selection of study participants will be depending on their health status and the investigators will exclude pediatric participants. Two blood samples will be collected from participants. First one is after the insertion of the intravenous peripheral line. The second is after fluid infusion through the same line. Samples will be sent to the laboratory then. Results will be collected and analyzed.

The importance of the research: If this type of sampling can be standardized , this means there will be less insertions to the patients, less adverse effects in relation to the number of insertions, fast and preexisted intravascular access for sampling so the time can be saved in critical conditions.

ELIGIBILITY:
Inclusion Criteria:

* It will include healthy adult volunteers.

Exclusion Criteria:

* Pediatric patients and critically ill patients will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of pCO2, pO2 (mmHg) Before and After IV Fluid Infusion in Healthy Adults | 1 year
  Blood samples will be analyzed using a venous blood gas (VBG) machine to assess pCO2, pO2 (mmHg). We will measure these values both before and after IVF infusion. The comparison of results aims to detect any statistically significant changes. This approach prioritizes patient comfort by utilizing the same catheter and requiring only a minimal blood discard.
Comparison of PH Before and After IV Fluid Infusion in Healthy Adults | 1 year
  Blood samples will be analyzed using a venous blood gas (VBG) machine to assess PH. We will measure these values both before and after IVF infusion. The comparison of results aims to detect any statistically significant changes. This approach prioritizes patient comfort by utilizing the same catheter and requiring only a minimal blood discard.
Comparison of ctHb (g/dL) Before and After IV Fluid Infusion in Healthy Adults | 1 year
  Blood samples will be analyzed using a venous blood gas (VBG) machine to assess ctHb (g/dL) . We will measure these values both before and after IVF infusion. The comparison of results aims to detect any statistically significant changes. This approach prioritizes patient comfort by utilizing the same catheter and requiring only a minimal blood discard.
Comparison of SO2, FO2Hb, FCOHb, FMetHb (%) Before and After IV Fluid Infusion in Healthy Adults | 1 year
  Blood samples will be analyzed using a venous blood gas (VBG) machine to assess SO2, FO2Hb, FCOHb, FMetHb (%). We will measure these values both before and after IVF infusion. The comparison of results aims to detect any statistically significant changes. This approach prioritizes patient comfort by utilizing the same catheter and requiring only a minimal blood discard.
Comparison of cBase(Ecf)c, cHCO,-(P.st)c, cNa, cK, cCl, cCa (mmol/L) Before and After IV Fluid Infusion in Healthy Adults | 1 year
  Blood samples will be analyzed using a venous blood gas (VBG) machine to assess cBase(Ecf)c, cHCO,-(P.st)c, cNa, cK, cCl, cCa (mmol/L). We will measure these values both before and after IVF infusion. The comparison of results aims to detect any statistically significant changes. This approach prioritizes patient comfort by utilizing the same catheter and requiring only a minimal blood discard.

CONTACTS AND LOCATIONS:
Overall Officials: Dunya N Alfaraj, MD, Principal Investigator — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Fahd University Hospital, Khobar, East, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Not decided yet